CLINICAL TRIAL: NCT05486065
Title: Investigation of Once-weekly Semaglutide S.C. Dose-Response in Patients With Type 2 Diabetes and Overweight - a Participant- and Investigator-blinded and Sponsor Open-label Study
Brief Title: A Research Study to Look Into How Well Semaglutide Medicine Works at Different Doses in People With Type 2 Diabetes and Overweight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-4984; U1111-1271-9209 (Other: World Health Organization (WHO)); 2022-000882-41 (EudraCT Number)
Record Dates: First submitted 2022-07-31; First posted 2022-08-03 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Semaglutide 2 mg (Experimental): Participants will receive once-weekly semaglutide 2 mg subcutaneous (s.c.) injection.
  Interventions: Drug: Semaglutide
- Semaglutide placebo 2 mg (Placebo Comparator): Participants will receive once-weekly semaglutide placebo 2 mg s.c. injection.
  Interventions: Drug: Placebo
- Semaglutide 8 mg (Experimental): Participants will receive once-weekly semaglutide 8 mg s.c. injection.
  Interventions: Drug: Semaglutide
- Semaglutide placebo 8 mg (Placebo Comparator): Participants will receive once-weekly semaglutide placebo 8 mg s.c. injection.
  Interventions: Drug: Placebo
- Semaglutide 16 mg (Experimental): Participants will receive once-weekly semaglutide 16 mg s.c. injection.
  Interventions: Drug: Semaglutide
- Semaglutide placebo 16 mg (Placebo Comparator): Participants will receive once-weekly semaglutide placebo 16 mg s.c. injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide s.c. injection once-weekly for 40 weeks. Dose gradually increased over 24 weeks, followed by a 16 week maintenance period.
  Arms: Semaglutide 16 mg; Semaglutide 2 mg; Semaglutide 8 mg
Drug: Placebo — Semaglutide placebo s.c. injection once-weekly for 40 weeks. Dose gradually increased over 24 weeks, followed by a 16 week maintenance period.
  Arms: Semaglutide placebo 16 mg; Semaglutide placebo 2 mg; Semaglutide placebo 8 mg

SUMMARY:
This study compares how three doses of semaglutide work in participants with type 2 diabetes (T2D) and overweight who are taking metformin. The study will look mainly at how well participant's blood sugar and participant's body weight are controlled when they are taking the study medicine at different doses. Participants will either get semaglutide [2 milligrams (mg), 8 mg, or 16 mg] or semaglutide placebo (a dummy medicine). Participants will take the study medicine with an injection pen called NovoPen®4. The injection pen is a medical tool with a needle used to inject the study medicine under the skin. The study will last for about 52 weeks. Participants will have 13 clinic visits and 4 phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus greater than equal to (≥) 180 days prior to the day of screening.
* Glycosylated haemoglobin (HbA1c) of 7.0 - 10.5 percentage (%) [53 - 91 millimoles per mole (mmol/mol)] (both inclusive).
* Body Mass Index (BMI) ≥ 27.0 kilograms per meter square (kg/m^2).
* Stable daily dose(s) ≥ 90 days prior to the day of screening of any metformin formulations.

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to day of screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of less than (<) 30 milliliters per minute (mL/min)/1.73 meter square (m^2) at screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (130):
- United States (101):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - University of Alabama Birmingham, Birmingham, Alabama
  - Velocity Clinical Res-Banning, Banning, California
  - Velocity Clin Res-Chula Vista, Chula Vista, California
  - Southern California Res Ctr, Coronado, California
  - Cedars-Sinai Medical Group, Encino, California
  - Velocity Clin Res Gardena, Gardena, California
  - Nat Res Inst Huntington Park, Huntington Park, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - First Valley Med Grp Lancaster, Lancaster, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Diabetes Assoc. Med Group, Orange, California
  - Western University of Health Sciences, Pomona, California
  - San Diego Family Care_San Diego, San Diego, California
  - Mills-Peninsula Hlth Services, San Mateo, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Optumcare Clinical Trials,LLC-Golden, Colorado Springs, Colorado
  - Innovative Research of W FL, Clearwater, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Alliance for Multispec Res, Coral Gables, Florida
  - University Clin Res-Deland, DeLand, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Indago Research & Health Center Inc., Hialeah, Florida
  - Northeast Res Inst. Inc., Jacksonville, Florida
  - New Life Medical, Miami, Florida
  - Genesis Research Center, LLC, Miami, Florida
  - Suncoast Clinical Research, Inc., Miami, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - San Marcus Res Clin Miami Lakes, Miami Lakes, Florida
  - Clinical Neuroscience Solution, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Family Clinical Trials, Pembroke Pines, Florida
  - Northeast Research Institute, Saint Augustine, Florida
  - St Johns Center for Clin. Res, Saint Augustine, Florida
  - Appalachian Clinical Res LLC, Adairsville, Georgia
  - Urban Family Practice Assoc, Marietta, Georgia
  - Herman Clinical Research LLC, Suwanee, Georgia
  - Rocky Mt Clin Res, LLC, Idaho Falls, Idaho
  - Velocity Clinical Res Boise, Meridian, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Biofortis Clinical Research, Addison, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - West Broadway Clinic, Council Bluffs, Iowa
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Norton Healthcare Research Office, Louisville, Kentucky
  - Barnum Medical Research Inc., Natchitoches, Louisiana
  - MedStar Community Clin Res Ctr, Hyattsville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Endo And Metab Cons, Rockville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Aa Mrc Llc, Flint, Michigan
  - Elite Research Center, Flint, Michigan
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - Arcturus Healthcare, PLC, Troy, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Premier Research Inc., Trenton, New Jersey
  - AMC Community Endocrinology, Albany, New York
  - Mid Hudson Med Res-New Windsor, New Windsor, New York
  - Northport VA Med Ctr Northport, Northport, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - UNC Eastowne Clinical Research Unit, Chapel Hill, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Providence Health Partners Ctr, Dayton, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - Velocity Clin Res Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Res Medford, Medford, Oregon
  - Lycoming Internal Medicine, Inc., Jersey Shore, Pennsylvania
  - Thomas Jefferson Univ Di Rsrch Ctr, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - CORE - Temple University, Philadelphia, Pennsylvania
  - Tower Health, West Reading, Pennsylvania
  - Velocity Clinical Research Columbia, Columbia, South Carolina
  - Velocity Clinical Research Greenville, Greenville, South Carolina
  - Coastal Carolina Res Ctr, Mt. Pleasant, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Velocity Clinical Research Union, Union, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Murphy Research Center, Humboldt, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Quality Research Inc, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - DCT-Stone Oak, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Dwayne O. Williams, M.D., P.A., Sugar Land, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Nova Health Management & Research Group, PC, Herndon, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Amherst Family Practice P.C., Winchester, Virginia
  - Velocity Clinical Research Spokane, Spokane, Washington
  - St. Vincent Hosp-Prevea Health, Green Bay, Wisconsin
  - Clinical Investigation Spec. Kenosha, Kenosha, Wisconsin
- Greece (12):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - Iatriko Psychicou Private Clinic, Athens
  - Gen Hospital of Athens Laiko,1st Dpt. of Propaedeutic Inter, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - Univ Gen Hospital Larisa, Larissa
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
- Hungary (8):
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged, Csongrád-Csanád
  - Komáromi Selye János Kórház, Komárom, Komárom-Esztergom
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - MH Egészségügyi Központ, Budapest
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Vas Vármegyei Markusovszky Egyetemi Oktatókórház, Szombathely
- Poland (8):
  - NBR Polska, Warsaw, Masovian Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - Ko-Med Centra Kliniczne Staszow, Staszów
  - NBR Polska Tomasz Klodawski, Warsaw
  - Clinmedica Research sp. z o.o., Skierniewice, Łódź Voivodeship
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Manati Ctr For Clin Research, Manatí, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 82 active sites in 4 countries, of which 75 sites enrolled participants.
Pre-assignment Details: Participants were randomized at a ratio of 3:1:3:1:3:1 to receive semaglutide (2 milligram [mg], 8 mg, 16 mg) or matching placebo.
Groups:
- Semaglutide 2.0 mg: Participants received once-weekly subcutaneous (s.c.) injections of semaglutide (in a dose-escalation manner every 4 weeks [0-4 weeks: 0.29 mg; 5-8 weeks: 0.58 mg; 9-12 weeks: 1.06 mg], followed by the maintenance dose of 2 mg) till 40 weeks.
- Semaglutide 8.0 mg: Participants received once-weekly s.c. injections of semaglutide (in a dose-escalation manner every 4 weeks [0-4 weeks: 0.29 mg; 5-8 weeks: 0.58 mg; 9-12 weeks: 1.06 mg; 13-16 weeks: 2.02 mg; 17-20 weeks: 4.03 mg], followed by the maintenance dose of 8 mg) till 40 weeks.
- Semaglutide 16.0 mg: Participants received once-weekly s.c. injections of semaglutide (in a dose-escalation manner every 4 weeks [0-4 weeks: 0.29 mg; 5-8 weeks: 0.58 mg; 9-12 weeks: 1.06 mg; 13-16 weeks: 2.02 mg; 17-20 weeks: 4.03 mg; 21-24 weeks: 8.06 mg], followed by the maintenance dose of 16 mg) till 40 weeks.
- Placebo: Participants received once-weekly s.c. injection of placebo matched to semaglutide for 40 weeks.
Period: Overall Study
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo
Started | 61 | 62 | 62 | 60
Full Analysis Set | 61 | 62 | 62 | 60
Safety Analysis Set | 60 | 60 | 62 | 59
Completed | 56 | 54 | 55 | 54
Not Completed | 5 | 8 | 7 | 6
Not completed — Withdrawal by Subject | 1 | 5 | 4 | 3
Not completed — Lost to Follow-up | 4 | 2 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Failure to meet randomization criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo | Total
Number analyzed (Participants) | 61 | 62 | 62 | 60 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (7.6) | 53.7 (7.5) | 52.9 (8.6) | 52.1 (9.5) | 52.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 25 | 35 | 120
  Male | 34 | 29 | 37 | 25 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 9 | 13 | 39
  Not Hispanic or Latino | 52 | 54 | 53 | 47 | 206
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 11 | 4 | 4 | 25
  White | 54 | 49 | 56 | 55 | 214
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to end of treatment (week 40) is presented.
Time Frame: Baseline (week 0) and End of treatment (week 40)
Population: Full analysis set included all randomised participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage-point of HbA1c
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 56 | 54
Percentage-point of HbA1c | -1.9 (1.1) | -1.8 (1.5) | -2.1 (1.5) | -1.1 (1.3)
Statistical Analysis 1: Comparison: Semaglutide 2.0 mg vs Placebo; Test type: Superiority — The change in HbA1c from baseline was analysed using an ANCOVA (Analysis of Covariance) with randomised treatment and stratification factor, sex as fixed effect and baseline HbA1c as a covariate. Missing values were imputed using Jump to reference method; p = 0.0002, ANCOVA; Treatment difference = -0.82, 95% CI 2-sided [-1.25 to -0.39]
Statistical Analysis 2: Comparison: Semaglutide 8.0 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0003, ANCOVA; Treatment difference = -0.77, 95% CI 2-sided [-1.19 to -0.35]
Statistical Analysis 3: Comparison: Semaglutide 16.0 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < .0001, ANCOVA; Treatment difference = -1.07, 95% CI 2-sided [-1.50 to -0.64]
Statistical Analysis 4: Comparison: Semaglutide 2.0 mg vs Semaglutide 8.0 mg; The change in HbA1c from baseline was analysed using an ANCOVA (Analysis of Covariance) with randomised treatment and stratification factor, sex as fixed effect and baseline HbA1c as a covariate. Missing values were imputed using Jump to reference method; Test type: Other; p = 0.8305, ANCOVA; Treatment difference = 0.05, 95% CI 2-sided [-0.38 to 0.47]
Statistical Analysis 5: Comparison: Semaglutide 8.0 mg vs Semaglutide 16.0 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1678, ANCOVA; Treatment difference = -0.30, 95% CI 2-sided [-0.72 to 0.13]
Statistical Analysis 6: Comparison: Semaglutide 2.0 mg vs Semaglutide 16.0 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2445, ANCOVA; Treatment difference = -0.25, 95% CI 2-sided [-0.67 to 0.17]

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to end of treatment (week 40) is presented.
Time Frame: Baseline (week 0) and End of treatment (week 40)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo
Number analyzed (Participants) | 56 | 56 | 55 | 53
Kilogram (kg) | -8.9 (8.5) | -10.1 (7.4) | -13.1 (8.4) | -2.3 (4.9)

3. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant that is temporally associated with use of investigational medicinal products (IMP), whether or not considered related to IMP. AE can therefore be any unfavourable & unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with use of IMP. TEAE was defined as event that had onset date (or increase in severity) during on-treatment observation period. On treatment observation period data are presented. On-treatment observation period is defined as time points from first drug date until first date of end of data point sets (DPS1) or last administration of randomised treatment +63 days. DPS1 in trial is defined as all observed data points from randomisation until first date of end of study visit or date of death or date of withdrawal of informed consent or contact as defined by investigator for participants that are lost to follow up.
Time Frame: From baseline (week 0) up to end of study (week 49)
Population: Safety analysis set included all participants who are exposed to randomised treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo
Number analyzed (Participants) | 60 | 60 | 62 | 59
Events | 43 | 54 | 55 | 37

4. Secondary Outcome: Number of Treatment-emergent Severe Hypoglycaemic Episodes
Description: Number of treatment-emergent severe Hypoglycaemic episodes are presented. Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. On treatment observation period data are presented. On-treatment oberservation period is defined as time points from first drug date until the first date of end of data point sets (DPS1) or last administration of randomised treatment +63 days. DPS1 in trial is defined as all observed data points from randomisation until the first date of end of study visit or date of death or date of withdrawal of informed consent or date of last contact as defined by investigator for participants that are lost to follow up.
Time Frame: From baseline (week 0) up to end of study (week 49)
Population: Safety analysis set included all participants who are exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo
Number analyzed (Participants) | 60 | 60 | 62 | 59
Episodes | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline (week 0) up to end of study (week 49)
Description: AEs presented here are TEAEs. TEAE was defined as event that had onset date (or increase in severity) during on-treatment observation period. On-treatment oberservation period define as time points from first drug date until the first date of end of data point sets (DPS1) or last administration of randomised treatment +63 days. Safety analysis set included all participants who are exposed to randomised treatment.
Arm/Group | Semaglutide 2.0 mg | Semaglutide 8.0 mg | Semaglutide 16.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/62 | 0/59
Serious Adverse Events (participants affected / at risk) | 4/60 | 2/60 | 1/62 | 2/59
Other Adverse Events (participants affected / at risk) | 30/60 | 48/60 | 50/62 | 29/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.0 mg (N=60) | Semaglutide 8.0 mg (N=60) | Semaglutide 16.0 mg (N=62) | Placebo (N=59)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.0 mg (N=60) | Semaglutide 8.0 mg (N=60) | Semaglutide 16.0 mg (N=62) | Placebo (N=59)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 4 (4) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 5 (6) | 2 (3) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (7) | 2 (4)
COVID-19 (Infections and infestations) | 1 (1) | 8 (8) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 8 (11) | 12 (16) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (29) | 20 (30) | 13 (19) | 7 (56)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6) | 3 (3) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 5 (5) | 5 (13) | 1 (1)
Eructation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (8) | 1 (2)
Fatigue (General disorders) | 2 (3) | 4 (4) | 6 (7) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (6) | 6 (13) | 7 (9) | 8 (23)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 3 (3) | 2 (2) | 3 (3) | 1 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 1 (1) | 3 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 13 (17) | 25 (54) | 23 (29) | 9 (18)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (16) | 14 (26) | 16 (32) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT05486065/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT05486065/SAP_001.pdf